CLINICAL TRIAL: NCT05789264
Title: Feasibility Study of a Nasal Compression Device in Comparison to Digital Nasal Compression for Stopping Epistaxis
Brief Title: Nasal Compression Device Study for Epistaxis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NasaClip (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMI001
Record Dates: First submitted 2023-02-26; First posted 2023-03-29 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Epistaxis Nosebleed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Participants assigned to the standard of care arm will be guided through clearing out clots in the nose (if using oxymetazoline), correct head positioning and how to appropriately hold nasal pressure and +/- oxymetazoline applied by a trained medical provider. No packing material will be inserted into the nares and only external pressure will be applied.
  Interventions: Diagnostic Test: Routine Care
- Nasal Compression Device (Experimental): Participants assigned to the nasal compression device arm will be provided with the device package which will include the compression device, nasal sponges, and +/- oxymetazoline nasal spray to apply to the sponges as well as written/graphical assembly and application instructions. Participants will then assemble and apply the device themselves under the supervision of a trained medical provider.
  Interventions: Device: Nasal Compression Device

INTERVENTIONS:
Device: Nasal Compression Device — Participants assigned to the NasaClip arm will not receive routine care as the objective of this study is to compare the NasaClip device to routine digital compression in terms of feasibility, comfort, and efficacy. Limited data previously discussed in the background section indicates that application of nasal compression devices may be superior to digital compression.
  Arms: Nasal Compression Device
Diagnostic Test: Routine Care — Most first aid instructions for epistaxis management tell patients to apply firm digital pressure for 10 to 20 minutes, use a topical vasoconstrictor and apply an ice pack over the nose.
  Arms: Standard of Care

SUMMARY:
This study will explore how a nasal compression device compares to manual compression for stopping anterior nosebleeds. This will be a non-randomized controlled trial enrolling participants presenting to medical care for anterior nosebleeds. Participants will be assigned to receive either a nasal compression device or standard of care consisting of digital compression. Participants will be asked to complete survey questions to assess satisfaction with the care they received, comfort, and overall experience with the device.

DETAILED DESCRIPTION:
This will be a non-randomized controlled trial study design. Alternating assignments will be made to either the nasal compression device arm or standard of care (manual nasal compression with pinching) arm.

Patients with anterior nosebleeds and not meeting any exclusion criteria will be identified upon registration at the study locations. The patient will be approached by a study team member who will briefly inform the patient about the study and invite the patient to participate. If the patient agrees to participate, they will be assigned to either the nasal compression device arm or the standard of care arm. Participants will then undergo a brief medical screening by a medical provider during the triage process to ensure no exclusion criteria are present. A study information sheet including key information, risks and benefits, and study team contact information will be provided for the patient to review while they are receiving treatment. Patients will be allowed to end their participation in the study at any time.

Participants will then be assessed every 5-10 minutes by a study team member to evaluate if bleeding has resolved. If a participant is still bleeding during a bleeding check they will be supplied a new device/gauze to avoid having to reuse bloodied material.

If bleeding has not resolved after 30 minutes of wearing the nasal compression device or with digital pressure, this will be defined as a treatment failure and patients will receive second line therapies at the discretion of the medical provider. Participants in the device arm will be provided with a NasaClip device upon discharge from the study site and all participants will be contacted 48 hours later to determine if they had further epistaxis at home, whether they used the device if given one, ease of application at home, and whether it was successful.

ELIGIBILITY:
INCLUSION

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Presenting with anterior epistaxis determined as someone with venous bleeding that can be controlled with external compression.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged at least 18.
4. In good general health as determined by the PI or Sub-I(s).

EXCLUSION

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Known allergic or hypersensitivity reactions to components of NasaClip or oxymetazoline.
2. Less than 18 years of age.
3. Known pregnancy.
4. Unable to provide informed consent.
5. Subjects who are prisoners or who are in police custody.
6. Identified by the medical team as having an acute exacerbation or poor control of any of the following medical conditions: high blood pressure, heart disease, thyroid disease, diabetes, trouble urinating due to an enlarged prostate.
7. Patients taking MAO inhibitors.
8. Medical instability or need for emergent intervention as determined by on-site medical team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome - Change over time from full epistaxis to cessation. | Checked at 10 min intervals for a total of 3 intervals (30 min).
  Primary outcome is time to bleeding cessation.

CONTACTS AND LOCATIONS:
Locations (1):
- Next Level Urgent Care, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Traboulsi H, Alam E, Hadi U. Changing Trends in the Management of Epistaxis. Int J Otolaryngol. 2015;2015:263987. doi: 10.1155/2015/263987. Epub 2015 Aug 16. PMID 26351457
- [Background] Bequignon E, Teissier N, Gauthier A, Brugel L, De Kermadec H, Coste A, Pruliere-Escabasse V. Emergency Department care of childhood epistaxis. Emerg Med J. 2017 Aug;34(8):543-548. doi: 10.1136/emermed-2015-205528. Epub 2016 Aug 19. PMID 27542804
- [Background] Padgham N. Epistaxis: anatomical and clinical correlates. J Laryngol Otol. 1990 Apr;104(4):308-11. doi: 10.1017/s0022215100112563. PMID 2370452
- [Background] Guarisco JL, Graham HD 3rd. Epistaxis in children: causes, diagnosis, and treatment. Ear Nose Throat J. 1989 Jul;68(7):522, 528-30, 532 passim. PMID 2676467
- [Background] Gifford TO, Orlandi RR. Epistaxis. Otolaryngol Clin North Am. 2008 Jun;41(3):525-36, viii. doi: 10.1016/j.otc.2008.01.003. PMID 18435996
- [Background] Schlosser RJ. Clinical practice. Epistaxis. N Engl J Med. 2009 Feb 19;360(8):784-9. doi: 10.1056/NEJMcp0807078. No abstract available. PMID 19228621
- [Background] Bende M, Loth S. Vascular effects of topical oxymetazoline on human nasal mucosa. J Laryngol Otol. 1986 Mar;100(3):285-8. doi: 10.1017/s0022215100099151. PMID 3950497
- [Background] Kucik CJ, Clenney T. Management of epistaxis. Am Fam Physician. 2005 Jan 15;71(2):305-11. PMID 15686301
- [Background] Tunkel DE, Anne S, Payne SC, Ishman SL, Rosenfeld RM, Abramson PJ, Alikhaani JD, Benoit MM, Bercovitz RS, Brown MD, Chernobilsky B, Feldstein DA, Hackell JM, Holbrook EH, Holdsworth SM, Lin KW, Lind MM, Poetker DM, Riley CA, Schneider JS, Seidman MD, Vadlamudi V, Valdez TA, Nnacheta LC, Monjur TM. Clinical Practice Guideline: Nosebleed (Epistaxis). Otolaryngol Head Neck Surg. 2020 Jan;162(1_suppl):S1-S38. doi: 10.1177/0194599819890327. PMID 31910111
- [Background] Doo G, Johnson DS. Oxymetazoline in the treatment of posterior epistaxis. Hawaii Med J. 1999 Aug;58(8):210-2. PMID 10487000
- See also: Approach to the adult with epistaxis - UpToDate — https://www.uptodate.com/contents/approach-to-the-adult-with-epistaxis
- See also: Epistaxis: Practice Essentials, Anatomy, Pathophysiology — https://emedicine.medscape.com/article/863220-overview#a6